CLINICAL TRIAL: NCT03160352
Title: Effects of a Virtual Reality-based Dual-task Exercise on Vestibular Function in Healthy Community Dwellers. A Pilot Study
Brief Title: Effects of Exergames on Vestibular Function in Healthy Community Dwellers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BASEC 2016-1220
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Vestibular Diseases
MeSH Terms: conditions — Vestibular Diseases | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exergame (Experimental): The Senso is a training system (dividat, Schindellegi, Switzerland) for improving physical and cognitive function was used as exergame. With foot pushes participants triggered on a pressure-sensitive plate. The Senso game was projected with a beamer at white wall. To promote head movement during training the direction of the beamer was vertical tilted (± 15°) and horizontal turned (90°) with a remote controlled power panner.
  Interventions: Other: Exergame

INTERVENTIONS:
Other: Exergame — In total, 10 sessions were accomplished including baseline and post intervention measurements. The remaining eight exercise sessions lasted 40 minutes, with an actual training duration of 20 minutes. This resulted in a cumulative total intervention exercise time of 160 minutes.

SUMMARY:
The aim is to assess the effects of virtual reality-based intervention on vestibular functions in healthy community dwellers.

DETAILED DESCRIPTION:
Elderly usually experience an age-related type of vestibular disorder, which involves vertigo, dizziness and poor postural stability. These symptoms seem to contribute to the "geriatric syndrome", which describes a complex symptomatology. It usually has multiple causes and must be considered interdisciplinary. This study will only consider healthy elderly with an expected age-related degeneration of the vestibular system. In terms of restoring vestibular functioning, compensation can be classified into adaptation, substitution and habituation. Adaptation enhances the Vestibulo-ocular reflex, which is equivalent to restoration. Habituation on the other hand, accustoms the affected person to a conflicting situation, in order that the response of the Vestibulo-ocular reflex is avoided. Substitution is distinguished in literature between sensory and behavioral, in which the sensorial substitution transfers the importance given to proprioceptive and visual inputs and the behavioral substitution refers to avoidance strategies e.g. immobilization, increased blink reflex and prevention of head rotations. Slower gait speed may also be a method used by elderly for compensation during a task when the base of support is unstable. Considering recommendation future studies should incorporate examinations of functional gaze stability during typical daily tasks in more familiar settings as opposed to laboratory assessments. Increased head movement may disturb balance and the risk of falling may be raised while walking stairs. As head stability is challenged during stair descent, elderly with age-related visual and vestibular impairment have problems with completing this quotidian task. A way to consider these observations in vestibular rehabilitation is the use of a virtual reality environment, which provides a motivating and pleasant method to train and that includes exercises requiring head turns. Successful use of virtual reality in rehabilitation of vestibular patients has previously been implemented. However, these studies did not particularly to exercise head turns by completing an orientation task.

ELIGIBILITY:
Inclusion Criteria:

Healthy community dwellers Adult male and female participant's (≥65 years) Signed informed consent after being informed

Exclusion Criteria:

Benign paroxysmal positional vertigo Acute pain Walking disability (independent walking <10 meters) Uncontrolled cardiovascular disease (e.g.: uncontrolled blood pressure) Weakness due to neurological problems

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2017-06-25 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Dynamic Visual Acuity (DVA) | 30 minutes
  The DVA is the measurement of visual acuity during head movement relative to baseline static visual acuity

SECONDARY OUTCOMES:
Functional Gait Assessment (FGA) | 15 minutes
  The FGA is used to measure disturbances in balance and gait
Extended Timed Get-Up-And-Go (ETGUG) | 15 minutes
  The time measured during each task and the overall time mirrors the functional mobility of the participant
Gait speed | 5 minutes
  Time was measured in with a stopwatch as the participants walked in the central 6 m of the walkway.
Simulator Sickness Questionnaire (SSQ) | 5 minutes
  The SSQ questionnaire assesses, cyber or virtual reality sickness

CONTACTS AND LOCATIONS:
Overall Officials: Swanenburg Jaap, PhD, Principal Investigator — University Hospital Zurich, Directorate of Research and Education, Physiotherapy & Occupational Therapy Research
Locations (1):
- University Hospital Zurich, Directorate of Research and Education, Physiotherapy & Occupational Therapy Research, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Publication

REFERENCES:
- [Derived] Swanenburg J, Wild K, Straumann D, de Bruin ED. Exergaming in a Moving Virtual World to Train Vestibular Functions and Gait; a Proof-of-Concept-Study With Older Adults. Front Physiol. 2018 Jul 31;9:988. doi: 10.3389/fphys.2018.00988. eCollection 2018. PMID 30108511